CLINICAL TRIAL: NCT00018473
Title: Gene-Environment Interactions in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: EPID-006-98F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Alzheimer's Disease
Keywords: Risk Factors; Genes; Epidemiology; Apolipoproteins E; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

SUMMARY:
This study will create Alzheimer 's disease risk profiles for defined combinations of genotypes and environmental exposures. This study will carry out a molecular epidemiologic study to identify genetic and environmental risks factors using state of the art techniques. The following will be done during the course of this study 1) Recruit both Alzheimer's patients and cognitively normal aged veterans. 2) Evaluate gene interaction in Alzheimer's disease. 3) Evaluate gene-environment interactions on the risk of Alzheimer's disease. These procedures should initially address the question as to whether certain genes either independently or synergistically modify the risk of Alzheimer's disease. This study will also determine whether certain environmental factors (smoking, alcohol consumption etc.) can modify the risk of AD and whether this effect is dependent on certain genetic backgrounds. This study will provide information that will be useful in designing therapies, develop risk factor profiles to be further tested in future studies, designating patients for specific therapies based on genetic factors and providing data and genetic material for future studies. This study will also provide a cohort of older and well characterized cognitively normal veterans for prospective genetic epidemiological studies on aging.

ELIGIBILITY:
The GRECC located at this hospital represents the leading edge of clinical care focusing on the needs of the aging veteran. We will recruit all 100 patients currently hospitalized at the Dementia Unit. We will also recruit from the outpatient memory clinic. We will enroll 400 AD patients total. Since, cases and controls will be ascertained from the same population, we also expect the socioeconomic status of individuals in these two groups to be the same. In the past year 9600 patients were treated on an outpatient basis. They were almost entirely white and male (>90%). The age demographics are 23% between 60-69, 23% between 70-79 and 5 % 80 or greater. The outpatients are seen for a wide variety of conditions. We plan to enroll 100 patients a year for 4 years (400 total). They will be seen once and have the same neuropsychological exams as the AD patients. Control subjects will be enrolled if their Mini-Mental score is greater than 24.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-04; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- VAMC- Bedford (Station 518), Bedford, Massachusetts, United States